CLINICAL TRIAL: NCT06170086
Title: Early Neurological Trajectory and Clinical Outcomes in Brain Acute Ischemic Stroke
Status: Active, not recruiting | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Xin Lou, Deputy Director of Department of Radiology, Chinese PLA General Hospital
Other Study IDs: brain acute ischemic stroke
Record Dates: First submitted 2023-12-06; First posted 2023-12-14 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Stroke, Acute
Keywords: Perforating artery; Acute stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective identification of potential responsible blood vessels, provision of intervention targets, prevention of fatal and disabling cerebrovascular diseases, identification of early END patients, determination of clinical treatment pathways, improvement of efficacy, and improvement of prognosis

DETAILED DESCRIPTION:
1. Research background： Stroke is divided into ischemic stroke and hemorrhagic stroke, with ischemic stroke accounting for about 70% and being the main type of stroke. The branch atherosclerotic disease (BAD) accounts for 10%~15% of all acute ischemic stroke (ALS), mainly involving lenticular artery (LSA), parapontine median artery (PPA), thalamic geniculate body artery, anterior choroidal artery Heubner's artery and thalamic perforating artery. Its clinical symptoms often manifest as early neurological deterioration (END), mainly progressive motor dysfunction (PDM), within 48 to 72 hours of onset, with an incidence rate of approximately 17% -75%. The clinical prognosis is poor.
2. The purpose and significance of the research Prospective identification of potential responsible blood vessels, provision of intervention targets, prevention of fatal and disabling cerebrovascular diseases, identification of early END patients, determination of clinical treatment pathways, improvement of efficacy, and improvement of prognosis
3. Research contents 1) Research on the relationship between stroke responsibility vessels and the pathogenesis of END in patients based on magnetic resonance three-dimensional time leap vascular imaging technology; 2) The impact of clinical interventions (intravenous thrombolysis, antiplatelet therapy, anticoagulation, statins, neuroprotective drugs, etc.) on END
4. Patient inclusion and exclusion criteria inclusion criteria

   1. Acute perforating atherosclerotic stroke patients within 48 hours of onset;
   2. Age ≥ 18 years and ≤ 80 years old;
   3. Having two or more vascular risk factors, including hypertension, diabetes, coronary heart disease, hyperlipidemia, smoking and obesity;
   4. Sign informed consent form exclusion criteria

   <!-- -->

   1. Patients with large artery stroke;
   2. Contraindications to magnetic resonance imaging or pregnant women;
   3. Other vascular lesions, such as aneurysms, vascular dissection, vasculitis, and brain tumors
5. Research method Select and treat emergency stroke patients according to the research design requirements, record clinical data, and evaluate the timing of 7T MRI. The patient underwent 7T MRI examination within 24 hours after the first diagnosis of acute stroke of the perforating artery, within 24 hours after aggravation, and 2 weeks after treatment according to the consensus of Chinese experts on perforating artery atherosclerosis. The sequences involved include: T1, T2flair, DWI, ADC, SWI, MRA, and high-resolution MRI of the responsible carrier artery (including cross section and longitudinal section). Collect original image images, search for the responsible perforating artery for stroke, calculate baseline core infarct volume (DWI), aggravated core infarct volume (DWI), and final infarct volume (T2 flair) after 2 weeks of treatment. Clinical evaluation baseline and NIHSS score after 3 months, to explore the relationship between responsible blood vessels and core infarct volume and NIHSS score.
6. Data statistical methods Measurement data that follow a normal distribution are expressed in the form of mean ± standard deviation, while non normal distribution measurement data are expressed in the form of median (25% percentile -75% percentile). Inter group comparison of econometric data with normal distribution and homogeneity of variance, using t-test or analysis of variance; The Wilcoxon rank sum test is used for inter group comparison of non normal distribution econometric data. The chi square test is used for inter group comparison of count data. Correlation analysis uses either Person correlation analysis or Spearman correlation analysis. The consistency test between methodologies was conducted using Kappa test.

ELIGIBILITY:
Inclusion Criteria:

A. Acute Perforating artery stroke patients within 48 hours of onset; B. Age ≥ 18 years and ≤ 80 years old; C. Have two or more vascular risk factors, including hypertension, diabetes, coronary heart disease, hyperlipidemia, smoking and obesity; D. Sign an informed consent form;

Exclusion Criteria:

A. Patients with large artery stroke; B. Contraindications to magnetic resonance imaging or pregnant women; C. Other vascular lesions, such as aneurysms, vascular dissection, vasculitis, and brain tumors;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A. Acute Perforating artery stroke patients within 48 hours of onset; B. Age ≥ 18 years and ≤ 80 years old; C. Have two or more vascular risk factors, including hypertension, diabetes, coronary heart disease, hyperlipidemia, smoking and obesity; D. Sign an informed consent form;
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Offending vessels | 5 years
  The blood vessels that cause stroke
Core infarct volume | 5 years
  The volume of high signal in the infarcted area on DWl or T2 FLAIR
NIH Stroke Scale (NIlSS） | 5 years
  The NIHSS score includes: consciousness level (consciousness level, consciousness level questioning, consciousness level instruction), gaze, field of vision, facial paralysis, upper limb movement, lower limb movement, limb ataxia, sensation, language, articulation disorders, and neglect. The scoring range is 0-42 points, with higher scores indicating more severe neurological damage

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China